CLINICAL TRIAL: NCT04843345
Title: A Prospective Cohort Study of Treatment Response in Sjogren's Syndrome-Related Lung Diseases Compared to Primary Idiopathic Lung Diseases
Brief Title: Sjogren's Lung Study
Status: Suspended | Type: Observational
Why Stopped: Indefinite paused for staffing issues
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jason Melehani, Clinical Fellow, Stanford University
Other Study IDs: IRB-59313
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Sjogren's Syndrome; Interstitial Lung Disease; Primary Pulmonary Lymphoma (Disorder); Chronic Bronchiolitis; Bronchiectasis; Lung Diseases; Cystic Lung Disease; Lymphocytic Interst. Pneumonitis
MeSH Terms: conditions — Sjogren's Syndrome; Lung Diseases, Interstitial; Bronchiectasis; Lung Diseases; Cystic Disease Of Lung; Lymphoid Interstitial Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reduced Salivary Flow Patients: Patients with lung disease matching inclusion criteria who screen positive for reduced salivary flow
- Normal Salivary Flow Patients: Patients with lung disease matching inclusion criteria who screen negative for reduced salivary flow

SUMMARY:
Lung involvement in Sjögren's syndrome is common and causes reduced quality of life and increased mortality. Sjögren's syndrome-related lung diseases (SS-RLD) are classified and treated as the primary lung diseases they resemble. Whether this approach is optimal has not been evaluated thoroughly. A critical gap in knowledge is knowing whether SS-RLDs have a unique clinical course and response to therapy. Given the underlying immune system dysfunction in Sjögren's syndrome, the investigators hypothesize that patients with SS-RLD will be more likely to respond to immunosuppressive therapy than patients with the matching primary lung disease. To address this hypothesis, the investigators will prospectively screen for Sjogren's syndrome in patients presenting to pulmonary clinics and compare the clinical course and response to therapy in Sjogren's syndrome positive and negative patients.

DETAILED DESCRIPTION:
Sjögren's syndrome is an autoimmune disease affecting at least 1% of adults characterized by hyperactive lymphocytes that damage exocrine glands leading to dry eyes and dry mouth. Although less well recognized, lung involvement in Sjögren's syndrome is common and causes reduced health-related quality of life and increased mortality. Sjögren's syndrome-related lung diseases are classified and treated as the primary lung diseases they resemble. Whether this approach is optimal has not been evaluated thoroughly.

Despite the potentially life-threatening consequence of Sjögren's syndrome-related lung disease, general medical education still promotes the false idea that Sjögren's syndrome is a nuisance disease. This leads many clinicians to overlook Sjögren's syndrome as a possible cause for respiratory symptoms. Even when Sjögren's syndrome is identified, there is no standard for attribution of the lung disease and little data on how to best treat it.

Only one study has compared interstitial lung disease patients with and without Sjögren's syndrome. Although it was a small retrospective study, it found that patients with usual interstitial pneumonia and Sjögren's syndrome were more likely to achieve stable lung function with immunosuppressive therapy as compared to the idiopathic cohort. This is striking as usual interstitial pneumonia is generally thought to not be responsive to immunosuppressive therapy.

A critical gap in knowledge is knowing whether Sjögren's syndrome-related lung diseases have a unique clinical course and response to therapy. Given the underlying immune system dysfunction in Sjögren's syndrome, the investigators hypothesize that patients with Sjögren's syndrome-related lung disease will be more likely to respond to immunosuppressive therapy than patients with the matching primary lung disease.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Interstitial Lung Disease and Other Parenchymal Lung Diseases

* Known or suspected interstitial lung disease regardless of radiographic pattern
* Interstitial lung disease due to alternative autoimmune etiology
* Sarcoidosis
* Organizing pneumonia
* Hypersensitivity pneumonitis absent known or suspected trigger
* Primary pulmonary lymphoma
* Other idiopathic pulmonary conditions at discretion of study team

Group 2: Refractory Airway Symptoms

* Chronic cough despite treatment trials with albuterol, proton-pump inhibitors and anti-histamine and intranasal corticosteroids
* Persistent bronchial hyperreactivity (defined as positive response to methacholine challenge on spirometry or subjective worsening after exposure to airway irritants such as tobacco, pollution, etc) or persistent asthma symptoms despite trial of inhaled corticosteroid and long acting bronchodilator
* Unexplained persistent bronchial wall thickening on CT imaging
* Recurrent or chronic bronchiolitis (including but not limited to chronic bronchiolitis, obliterative bronchiolitis, lymphocytic bronchiolitis, constrictive bronchiolitis associated with bronchiolar destruction, and panbronchiolitis)
* Bronchiectasis
* Lymphocytic alveolitis on bronchoalveolar lavage absent hypersensitivity pneumonitis with known trigger or HIV
* Recurrent bacterial pneumonia (greater than 2 episodes in 1 year, confirmed by focal consolidative opacity on chest imaging and requiring antibiotic therapy)

Group 3: Other

•Select patients outside the protocol testing schema who have one of the above lung diseases and are found to have Sjogren's syndrome through the course of their normal clinical care will be invited to participate in the data collection portion of the study for analyzing longitudinal outcomes.

Exclusion Criteria:

* Patients with interstitial lung disease due to a known or suspected trigger such as drug-induced (including but not limited to nitrofurantoin, amiodarone, methotrexate and other chemotherapies), inorganic dust exposure (including but not limited to asbestos, silica, hard metals, coal dust) or organic exposure (including but not limited to birds, hay, mold).
* Patients who have taken a muscarinic antagonist or agonists within 7 days of planned testing
* Patients who are unable to consent for themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators aim to capture a wide range of adult patients with lung disease to better understand the contribution of Sjogren's syndrome to lung disease
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary function over time | Change from first test after enrollment to final test across 5-year monitoring period
  Based on underlying lung disease, standard measures of lung function (FEV1 vs FVC) will be followed

SECONDARY OUTCOMES:
Annual rate of hospitalizations from respiratory cause | Over 5-year monitoring period
Percent of participants who die from respiratory cause | Over 5-year monitoring period

CONTACTS AND LOCATIONS:
Overall Officials: Jason H Melehani, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No